CLINICAL TRIAL: NCT05387837
Title: A 3 Stage Ph 2 Study: St 1: Single SubQ D-4517.2 Dose Safety and PD in Wet wAMD or DME. Stage 1A: Multiple SubQ D-4517.2 Dose Safety, PK and PD in wAMD and DME. Stage 2: Safety, Tolerability, PK and Efficacy of SubQ D-4517.2 in wAMD
Brief Title: Safety, Tolerability and PK of Subcutaneous D-4517.2 in Subjects With Wet AMD or DME
Acronym: Tejas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ashvattha Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-4517-002
Record Dates: First submitted 2022-05-13; First posted 2022-05-24 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Stage 1 wAMD (Experimental): * Cohort A1 - 0.18 mg/kg of D-4517.2
  * Cohort B1 - 0.36 mg/kg of D-4517.2
  * Cohort C1 - 0.71 mg/kg of D-4517.2
  * Cohort D1 - 1.5 mg/kg of D-4517.2
  Interventions: Drug: D-4517.2
- Stage 1 DME (Experimental): * Cohort B2 - 0.36 mg/kg of D-4517.2
  * Cohort C2 - 0.71 mg/kg of D-4517.2
  * Cohort D2 - 1.5 mg/kg of D-4517.2
  Interventions: Drug: D-4517.2
- Stage 1A wAMD (Experimental): * Cohort E1 - 2.0 mg/kg of D-4517.2 every 2 weeks
  * Cohort F1 - 2.0 mg/kg of D-4517.2 every 4 weeks
  Interventions: Drug: D-4517.2
- Stage 1A DME (Experimental): * Cohort E2 - 2.0 mg/kg of D-4517.2 every 2 weeks
  * Cohort F2 - 2.0 mg/kg of D-4517.2 every 4 weeks
  Interventions: Drug: D-4517.2

INTERVENTIONS:
Drug: D-4517.2 — D-4517.2 (hydroxyl dendrimer VEGFR tyrosine kinase inhibitor)
  Other Names: aflibercept

SUMMARY:
A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of D-4517.2 After Subcutaneous Administration in subjects with Neovascular (wet) Age-Related Macular Degeneration (AMD) or subjects with Diabetic Macular Edema (DME)

DETAILED DESCRIPTION:
A Three Stage Phase 2 Study: Stage 1: Single Subcutaneous Dose Open-Label Assessment of Safety and Pharmacodynamic Response to D-4517.2 (hydroxyl dendrimer VEGFR tyrosine kinase inhibitor) in Subjects with Neovascular (wet) Age-Related Macular Degeneration (wAMD) or Subjects with Diabetic Macular Edema (DME). Stage 1A: Multiple Subcutaneous Dose Open-Label Assessment of Safety, Pharmacokinetics and Pharmacodynamic Response to D-4517.2 Co-administered with Aflibercept in Subjects with wAMD and DME. Stage 2: Visual Examiner-Masked, Randomized Active, Sham and Placebo Controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of a Subcutaneously Administered D-4517.2 to Subjects with wAMD

ELIGIBILITY:
Target population:

Inclusion Criteria:

Overall Study Inclusion Criteria-For All Subjects:

1. Willing and able to give informed consent, comply with all study procedures, and be likely to complete the study.
2. Demonstrated response to prior anti-VEGF treatment as defined by one or more of the following and as assessed by the Investigator for Stages 1 and 1A and confirmed by the Central Reader for Stage 2:

   1. Complete resolution or partial reduction of foveal intra- and/or subretinal fluid ≥ 30% from initial diagnosis as measured by SD-OCT.
   2. Increase in BCVA ≥ 2 lines from initial diagnosis using Snellen scale.
3. Female subjects may be enrolled if they are:

   1. Not pregnant, lactating, or breastfeeding
   2. Documented in medical records or subject self-reported to be surgically sterile or postmenopausal.
   3. Female subjects of childbearing potential must practice true abstinence for at least 28 days prior to investigational product (IP) administration until 30 days after the last IP administration and have a negative serum and urine pregnancy test at Screening and Baseline Day 1, respectively, or
   4. Using 2 forms of highly effective contraception, including 1 physical barrier (condom or diaphragm) plus another method, such as adequate hormonal method (eg, contraceptive implants, injectables, or oral contraceptives) or nonhormonal methods (eg, intrauterine device or spermicidals) from Screening or at least 2 weeks prior to IP administration (whichever is earlier) until 30 days after the last IP administration and having a negative serum and urine pregnancy test at Screening and Baseline Day 1, respectively.
4. Male subjects with female partners of childbearing potential may be enrolled if they are:

   1. Documented to be surgically sterile (vasectomy) in medical records or subject self-reported, or
   2. Agree to practice true abstinence during the study and for 30 days after the last IP administration, or
   3. Agree to use 2 adequate forms of highly effective contraception during the study, 1 of which should be a physical barrier for 30 days after the last IP administration.
   4. Must agree not to donate sperm during study and for 30 days following administration of the last dose of IP.
5. Subjects who complete the Aflibercept Treatment Period in Stage 1 are eligible to enroll in Stage 1A if they meet all eligibility requirements. These subjects will enter the study in the D-4517.2 Treatment Period.
6. Subjects who complete Stage 1 and/or Stage 1A are eligible to enroll in Stage 2 if they meet all eligibility requirements.
7. Ocular media clarity, pupillary dilation and individual cooperation sufficient for adequate fundus imaging in the opinion of the Investigator.
8. Recurrence of intra- or subretinal fluid at study Baseline. This inclusion criterion will be confirmed by the Sponsor or Central Reader in Stages 1 and 1A and by the Central Reader in Stage 2.
9. For subjects with bilateral disease, only one eye per subject can participate in the study. In cases where both eyes are eligible, the eye with the worse BCVA at the Screening Visit will be selected as the study eye. If both eyes have the same BCVA, the eye with the largest CST will be selected as the study eye.

   Subjects With wAMD (For all Stages):
10. Male or nonpregnant female adults aged ≥50 years at time of signing the informed consent form (ICF).
11. BCVA letter score between 75 and 23 letters (ETDRS chart) (20/32 to 20/320 Snellen equivalents) inclusive in the study eye at Baseline and BCVA letter score of at least 35 letters (ETDRS chart) (20/200 Snellen equivalent) in the non-study eye.
12. Previously treated subjects with at least 3 prior IVT injections with an anti-VEGF agent (aflibercept, bevacizumab, faricimab, ranibizumab, or any other approved anti-VEGF agent) with last treatment administered between 4 and 12 weeks prior to Screening. Administration of IVT anti-VEGF agents prior to enrollment must not be more than 12 weeks apart. This inclusion criterion will be assessed by the Investigator.
13. For Stage 2, presence of a choroidal neovascular (CNV) lesion secondary to wAMD confirmed by the Central Reader.
14. The Investigator attributes the cause of the decreased vision in the study eye primarily to wAMD.

    Subjects With DME (For Stages 1 and 1A only):
15. Male or nonpregnant female adults aged ≥18 years at time of signing the ICF.
16. Diagnosis of diabetes mellitus (Type 1 or Type 2). Any of the following will be considered to be sufficient evidence that diabetes is present:

    1. Current regular use of oral anti-hyperglycemic agents for the treatment of diabetes.
    2. Current regular use of insulin or other injectable drugs (eg, dulaglutide and liraglutide) for the treatment of diabetes.
    3. Documented diabetes by American Diabetic Association (ADA) and/or World Health Organization (WHO) criteria.
17. Hemoglobin A1c (HbA1c) ≤12% at Screening.
18. DME defined as macular thickening involving the center of the macula with CST of ≥325 μm using Spectralis® (Heidelberg Engineering, Heidelberg, Germany) SD-OCT at Screening. These inclusion criteria will be assessed by the Central Reader.
19. BCVA letter score between 75 and 23 letters (ETDRS chart) (20/32 to 20/320 Snellen equivalents) inclusive in the study eye at Baseline.
20. Previously treated subjects with at least 5 prior IVT injections with an anti-VEGF agent (aflibercept, bevacizumab, faricimab, ranibizumab, or any other approved anti-VEGF agent) with last treatment administered between 4 and 12 weeks prior to Screening. Administration of IVT anti-VEGF agents prior to enrollment must not be more than 12 weeks apart. This inclusion criterion will be assessed by the Investigator.
21. The Investigator attributes the cause of the decreased vision in the study eye primarily to DME.

Exclusion Criteria:

A subject who meets any of the following exclusion criteria will not be eligible for inclusion in the study:

Medical Conditions:

1. History, within 6 months prior to Screening, of any of the following: myocardial infarction, any cardiac event requiring hospitalization, treatment for acute congestive heart failure, transient ischemic attack or stroke.
2. Uncontrolled hypertension with systolic BP ≥160 mmHg and/or diastolic BP ≥100 mmHg (while subject at rest) at the Screening Visit. If the subject's initial reading exceeds these values, a second reading may be taken 30 minutes later on the same day. If the subject's BP is controlled by antihypertensive medication, the subject should be taking the same medication continuously for at least 30 days prior to Day 1.
3. Currently untreated diabetes mellitus, uncontrolled diabetes mellitus defined as HbA1c > 12%, or previously untreated subjects with diabetes mellitus who initiated oral or injectable anti-diabetic medication within 3 months prior to Day 1.
4. Chronic renal disease requiring chronic hemodialysis or renal transplantation.
5. Abnormal liver function, as defined by transaminase or total bilirubin 2 times above the upper limit of normal at the Screening Visit.
6. Medical history of Wolff-Parkinson-White Syndrome, family history of long QT or planned initiation or currently on medication prolonging QT time during the trial.
7. Known allergy to constituents of the study drug formulation, aflibercept, or clinically relevant hypersensitivity to fluorescein used by the subject during the study.
8. Serious systemic infections:

   1. Any active infections for which systemic anti-infectives were used within 4 weeks before Screening Visit.
   2. Recurrent or chronic infections or other active infections that, in the opinion of the Investigator, might cause this study to be detrimental to the subject.
9. Any organic or psychiatric disorder, or laboratory abnormality which, in the opinion of the Investigator, will prevent the subject from completing the study activities as in the protocol or interfere with the interpretation of the study results.
10. An underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious, or gastrointestinal) or history of other disease, physical examination finding or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of study drug, might affect interpretation of the results of the study or which, in the opinion of the Investigator, renders the subject at unacceptable risk of treatment complications by participating in the trial.
11. Any major illness or surgical procedure within 1 month before Screening.
12. History of other diseases, physical examination finding, historical or current clinical laboratory finding giving reasonable suspicion of condition that contraindicates the use of the IP or that might affect the interpretation of the results of the study or renders the subject at high risk for treatment complications, in the opinion of the Investigator.
13. Positive screen antibodies for hepatitis B or hepatitis C virus subsequently confirmed to suggest active infection, or HIV type 1 or 2 antibodies.

    Prior/Concomitant Therapy:
14. Participation in any investigational study within 30 days prior to Screening, or planned use of an IP or device during the study; any exposure to a prior investigational drug product must be fully washed out (at least 5 half-lives).
15. Chronic alcohol or drug abuse or any condition that, in the Investigator's opinion, makes them an unreliable study participant or unlikely to complete the trial.
16. Use of systemic medications known to be toxic to the lens, retina or optic nerve (eg, deferoxamine, chloroquine/hydroxy-chloroquine, tamoxifen, phenothiazines, and ethambutol) used during the 6 month or 5 half-lives (whichever is longer) prior to Day 1 or likely need to be used.
17. Use of systemic immunomodulatory treatments (eg, interleukin-6 inhibitors) within 6 months or 5 half-lives (whichever is longer) prior to Day 1.
18. Use of systemic corticosteroids (ie, oral, IM, IV, intranasal) within 1 month prior to Day 1 and no corticosteroids anticipated throughout the trial.
19. Systemic treatment for suspected or active systemic infections.
20. Administration of systemic anti-VEGF or pro-VEGF treatment within 180 days or 5 half-lives, whichever is longer, before Screening Visit.
21. Received blood transfusion within 3 months prior to the Screening Visit.

    Ocular Exclusion Criteria For Study Eye:
22. High risk proliferative diabetic retinopathy (DR) as assessed by the Investigator.
23. Any history of or ongoing rubeosis iridis.
24. Prior macular photocoagulation (defined as ≥ 100 burns placed previously outside of the posterior pole) in the study eye prior to Screening or expected to be received between the Screening Visit and Day 1.
25. History of treatment with periocular or IVT corticosteroids in the study eye in the past 3 months and no such treatment planned for the time between Screening and Day 1.
26. Treatment of DME or DR with macular laser.
27. Any intraocular surgery (eg, Cataract surgery) performed within 3 months prior to Screening or planned during the trial in the study eye.
28. Spherical equivalent of the refractive error in the study eye demonstrating more than -8 diopters of myopia (prior to cataract or refractive surgery) at the Screening Visit.
29. Uncontrolled intraocular pressure (IOP), defined as an IOP ≥ 25 mmHg, despite antiglaucoma medications in the study eye(s) at the time of Screening or controlled glaucoma that requires management with >2 topical hypotensive medications.
30. Presence of any clinically significant epiretinal membrane or vitreomacular traction in the study eye(s).
31. History or evidence of any of the following surgeries or procedures in the study eye(s):

    1. Sub-macular surgery or other surgical intervention.
    2. Prior retinal detachment or macular hole interventions.
    3. History of vitreoretinal surgery or vitrectomy.
    4. Photodynamic therapy or thermal laser retinal treatment of the macula or fovea.
    5. Intraocular laser treatments for glaucoma (eg, selective laser trabeculoplasty or peripheral iridotomy).
    6. Glaucoma filtering surgery (eg, trabeculectomy) or glaucoma drainage device (eg, Ahmed valve or Baerveldt valve) including minimally invasive glaucoma shunts (eg, minimally invasive glaucoma surgery.
    7. Neodymium: yttrium-aluminum-garnet (Nd:YAG) laser capsulotomy within the 30 days prior to the Screening Visit.
    8. Corneal refractive procedures (laser-assisted in situ keratomileusis [LASIK] or photorefractive keratectomy) within the 6 months prior to the Screening Visit or planned during the study.
    9. Corneal transplantation surgery.
32. History or clinical evidence of other concurrent conditions deemed by the Investigator likely to impact the subject's clinical safety or interfere with interpretation of study results including, but not limited to:

    1. Inflammatory conditions of the anterior or posterior segment (eg, chronic keratoconjunctivitis, uveitis, retinal vasculitis, neuritis, iritis, scleritis, or blepharitis) in either eye.
    2. Subretinal hemorrhage that is ≥ 50% of the total CNV lesion area.
    3. Any vitreous opacity that prevents proper visualization of the fundus and/or adversely alters visual acuity, in the opinion of the Investigator.
    4. Prior radiation therapy in the region of the eyes.
33. Presence of fibrosis as measured by SD-OCT and assessed by the Central Reader in Stages 1 and 1A. Fibrosis or atrophy of more than 50% of the lesion size and/or involving the foveal center of the study eye at Screening; these criteria will be assessed by the Central Reader in Stage 2.
34. Current or history of vitreous hemorrhage in the study eye within 3 months of Screening.
35. Any history of active or suspected ocular or periocular bacterial, viral, fungal or parasitic infections (eg, infectious or noninfectious conjunctivitis, keratitis, scleritis, endophthalmitis or other) in either eye within 30 days prior to Screening Visit.

    Other:
36. Has any finding that, in the view of the Investigator or Medical Monitor, would compromise the subject's safety requirements.
37. Any previous treatment with ILUVIEN, Ozurdex, or Retisert (fluocinolone acetonide IVT implant) in the non-study eye.
38. DME subjects who have BCVA of hand motion or worse in the non-study eye or non-physical presence of a non-study eye (ie, monocular).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2025-05-09 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Stage 1 Safety Evaluation | 12 weeks
  Safety of single dose of D-4517.2 as measured by Treatment-Emergent Adverse Events (TEAEs)
Stage 1A Safety Evaluation | 40 Weeks
  Safety of multiple SC doses of D-4517.2 as measured by Treatment-Emergent Adverse Events (TEAEs)

SECONDARY OUTCOMES:
Stage 1: Number of participants with a reduction in sub-retinal fluid after a single intravitreal (IVT) dose of aflibercept and a single SC dose of D-4517.2 | Within subject, percent reduction in subretinal fluid volume in study eye after IVT aflibercept and D-4517.2 at 2, 4, 6, 8, and 12 weeks post-dose measured by spectral domain optical coherence tomography (SD-OCT).
  Change in sub-retinal fluid as measured by spectral domain optical coherence tomography (SD-OCT).
Stage 1: Number of participants with duration of effect of D-4517.2 as assessed by changes in subretinal fluid over time up to 12 weeks | Within subject, central subfield thickness (CST) in study eye after IVT aflibercept and D-4517.2 at 2, 4, 6, 8, and 12 weeks post-dose as assessed by SD-OCT.
  Effect of D-4517.2 as measured by spectral domain optical coherence tomography (SD-OCT).
Stage 1: Number of participants with Ocular and non-ocular adverse events (AEs) and serious adverse events (SAEs) observed for D-4517.2 and aflibercept | By dose level, mean difference in percent reduction in subretinal fluid in study eye after IVT aflibercept and D-4517.2 at 2, 4, 6, 8, and 12 weeks post-dose as measured by SD-OCT.
  Participants with ocular and non-ocular adverse events and serious adverse events as measured by CTCAE v5.0
Stage 1: Number of participants with change in best corrected visual acuity (BCVA) in study eye after each treatment (aflibercept or D-4517.2). | Change from baseline in BCVA in study eye as assessed by early treatment of diabetic retinopathy scale (ETDRS) after each treatment (aflibercept and D-4517.2) at 4, 6, 8, and 12 weeks post-dose.
  Participants with change in vision as measured best corrected visual acuity (BCVA) assessment.
Stage 1A: Effect of different D-4517.2 dose regimens to maintain BCVA and CST following a single IVT aflibercept dose | 12 weeks of Aflibercept and 40 weeks of D-4517.2
  Change from baseline in study eye BCVA measured by ETDRS letter score and in study eye CST and intra/sub-retinal fluid volume measured by SD-OCT
Stage 1A: Pharmacokinetics (Cmax) of D-4517.2 Repeat Dosing | 24 Weeks
  D-4517.2 Cmax over the course of the study with repeat dosing
Stage 1A: Pharmacokinetics (AUC) of D-4517.2 Repeat Dosing | 24 Weeks
  D-4517.2 AUC over the course of the study with repeat dosing
Stage 1A: Pharmacokinetics (Tmax) of D-4517.2 Repeat Dosing | 24 Weeks
  D-4517.2 Tmax over the course of the study with repeat dosing
Stage 1A: Pharmacokinetics (CL/F) of D-4517.2 Repeat Dosing | 24 Weeks
  D-4517.2 CL/F over the course of the study with repeat dosing
Stage 1A: Rescue Treatment | 12 weeks of Aflibercept and 40 weeks of D-4517.2
  Time in weeks for rescue treatment during each Treatment Period and proportion of treated subjects remaining rescue-free at each study visit

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Macro Trials, Los Angeles, California
  - University Retina - Lemont, Lemont, Illinois
  - Midwest Eye Institute - North, Indianapolis, Indiana
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Springield Clinic, Springfield, Missouri
  - The Retina Institute - Clayton Office, St Louis, Missouri
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Erie Retina Research, Eire, Pennsylvania
  - Texas Retina Associates - Arlington, Arlington, Texas
  - Austin Retina Associates, Austin, Texas
  - Medical Center Ophthalmology Associates - Northwest, San Antonio, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Strategic Clinical Research Group, Willow Park, Texas
  - Virginia Retina Center, Leesburg, Virginia
  - West Virginia University Eye Institute, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No